CLINICAL TRIAL: NCT06936579
Title: Cortical Effects of Peripheral Proprioceptive Stimulation on the Motor Evoked Potentials of the Limbs
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Facultat de ciencies de la Salut Universitat Ramon Llull (Other)
Responsible Party: Principal Investigator, Pedro Victor López Plaza, Principal Investigator,, Facultat de ciencies de la Salut Universitat Ramon Llull
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 2025-04-07
Record Dates: First submitted 2025-04-12; First posted 2025-04-20 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Healthy Subjects

STUDY DESIGN:
Intervention Model Description: Each participant will serve as their own control and will be assessed under both stimulation (experimental) and no-stimulation (control) conditions
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Condition without proprioceptive stimulation: (No Intervention): Participants will not receive the stimulus, and MEP activity will be recorded under the same motor cortex stimulation conditions.
- Condition with proprioceptive stimulation 1 (Experimental): Participants will receive proprioceptive stimulation through the output plunger, applied continuously for 15 seconds, with 20-second rest intervals, over a total duration of 5 minutes. MEP activity will then be recorded via motor cortex stimulation.
  Interventions: Device: proprioceptive stimulation
- Condition with proprioceptive stimulation 2 (Active Comparator): Participants will receive proprioceptive stimulation continuously during the application of TMS pulses while MEP activity is recorded.
  Interventions: Device: proprioceptive stimulation

INTERVENTIONS:
Device: proprioceptive stimulation — Condition without proprioceptive stimulation: Participants will not receive the stimulus, and MEP activity will be recorded under the same motor cortex stimulation conditions.
  Condition with proprioceptive stimulation 1: Participants will receive proprioceptive stimulation through the output plunger, applied continuously for 15 seconds, with 20-second rest intervals, over a total duration of 5 minutes. MEP activity will then be recorded via motor cortex stimulation.
  Condition with proprioceptive stimulation 2: Participants will receive proprioceptive stimulation continuously during the application of TMS pulses while MEP activity is recorded.
  Arms: Condition with proprioceptive stimulation 1; Condition with proprioceptive stimulation 2

SUMMARY:
Through motor muscle potentials, we will observe how a peripheral somatosensory mechanical stimulus on key limb musculature communicates signals via afferent sensory fibers that encode proprioceptive signals from muscle spindles (particularly type Ia fibers) to the somatosensory cortex at rest, confirming the integrative hypothesis of movement.

These results would support interventions aimed at addressing sensory deafferentation present in multiple health conditions related to movement disorders, where disuse or immobilization lead to changes in movement patterns and a decrease in neuronal activation in somatosensory cortex areas involved in constructing voluntary movement.

DETAILED DESCRIPTION:
Objective: To evaluate whether a proprioceptive stimulus applied to the limb of healthy subjects activates the corticospinal pathway, compared to a condition without stimulation, through the analysis of motor evoked potentials (MEPs).

Methods: Experimental and crossover. Each participant will serve as their own control and will be assessed under both stimulation (experimental) and no-stimulation (control) conditions.The stimulus will consist of intermittent mechanical pressure on the skin located at the neuromuscular motor points (NMPs) of the upper limb (biceps muscle (B) and wrist extensors (WE)) and the lower limb (rectus femoris of the quadriceps (RFQ) and tibialis anterior (TA).Motor evoked potentials (MEPs) will be recorded from the B, WE, RFQ, and TA muscles using transcranial magnetic stimulation (TMS).The optimal stimulation point (hotspot-the area where TMS generates the highest MEP) will be identified individually for the B, WE, RFQ, and TA muscles.Participants will be recruited at the facilities of the Faculty of Physiotherapy and Nursing of Castilla-La Mancha University (UCLM), in collaboration with the Toledo Physiotherapy Research Group (GIFTO) and the Faculty of Health Sciences, Blanquerna - Ramon Llull University.

ELIGIBILITY:
Inclusion Criteria:

Good health status with no history of neuromuscular injuries, surgical interventions, or trauma affecting the central or peripheral nervous system.

Not currently taking drugs or medications known to affect the central nervous system, and not pregnant at the time of testing.

No metallic or electronic implants and no history of epilepsy.

(Safety, ethical considerations, and application guidelines for the use of transcranial magnetic stimulation in clinical practice and research)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 31 (Estimated)
Dates: Start 2025-05-20 (Estimated); Primary Completion 2025-07-15 (Estimated); Study Completion 2025-07-30 (Estimated)

PRIMARY OUTCOMES:
Motor evoked potentials (MEPs) | 45 minuts
  transcranial magnetic stimulation (TMS)

CONTACTS AND LOCATIONS:
Locations (1):
- Pedro Victor López Plaza, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No